CLINICAL TRIAL: NCT03121144
Title: Usability Validation of Patient Monitoring Device for Pressure Injury Prevention and Fall Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RAMS0006
Record Dates: First submitted 2017-03-27; First posted 2017-04-19 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Pressure Ulcer; Pressure Injury; Falls Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Masimo Centroid System (Experimental): Single-arm study. All subjects are enrolled into the test group wherein the noninvasive positional monitoring device will be administered.
  Interventions: Device: Masimo Centroid System

INTERVENTIONS:
Device: Masimo Centroid System — Noninvasive positional monitoring device

SUMMARY:
This study describes a procedure to collect a subject's position, movement, physiological data and usability information using Masimo's investigational device.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. ICU patient
3. Primarily bedbound subjects
4. Able to be monitored for a minimum of approximately 8 hours

Exclusion Criteria:

1. Pregnancy
2. Prisoner status
3. Pressure injury stage 2, 3, or ungroupable
4. Has a pacemaker or internal defibrillator
5. Has a history of complications with a similar study
6. Has any medical condition which in the judgment of the Investigator, renders them inappropriate for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Masimo Centroid System: All subjects are enrolled into the test group wherein the noninvasive positional monitoring device will be administered.
Period: Overall Study
Arm/Group | Masimo Centroid System
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Masimo Centroid System
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 14
  Asian | 2
  Asian/Native Hawaiian | 1
  White | 17
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Usability Validation of Masimo Centroid System
Description: The number of participants enrolled to assess the usability of the Masimo Centroid System.
Time Frame: At least 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Masimo Centroid System
Number analyzed (Participants) | 34
Participants | 34

ADVERSE EVENTS:
Time Frame: at least 8 hours and up to 16 hours of enrollment.
Arm/Group | Masimo Centroid System
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03121144/Prot_SAP_000.pdf